CLINICAL TRIAL: NCT03561636
Title: Health Literacy in the General Population in Belgium: Associations and Determinants
Brief Title: Health Literacy in the General Population in Belgium
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Collaborators: Solidaris (Unknown)
Responsible Party: Principal Investigator, Isabelle Bragard, Lecturer, University of Liege
Other Study IDs: HL-Solidaris
Record Dates: First submitted 2018-05-23; First posted 2018-06-19 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Health Literacy
Keywords: Health literacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aims of the study are:

* To measure health literacy (HL) levels in a sample composed of members of a health mutual (Solidaris), and its potential associations with several determinants (health, health services consumption, health behaviours...)
* To identify potential groups at risk of a lower HL
* To identify the determinants of HL level

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* Affiliated to Solidaris (health mutual), with a valid phone number
* Consent to participate

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults affiliated to Solidaris
Sampling Method: Probability Sample
Enrollment: 2535 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Health Literacy | At the inclusion in the study
  The degree to which individuals can obtain, process and understand basic health information and services needed to make appropriate health decisions. It also includes the cognitive and social skills which determine the motivation and ability of individuals to gain access to, understand and use information in ways which promote and maintain good health. It is measured by the Health Literacy Questionnaire (HLQ) (Osborne et al., 2013), composed of 44 items (9 dimensions).

SECONDARY OUTCOMES:
General health | At the inclusion in the study
  Measured with the EQ-5D-5L (EuroQol Group, 1990), divided into 2 parts. The first part is composed of 5 items investigating 5 dimensions (mobility, autonomy, daily activities, pain, and anxiety and depression).
General health | At the inclusion in the study
  Measured with the EQ-5D-5L (EuroQol Group, 1990), divided into 2 parts: the second part is composed of 1 Visual Analogue Scale (VAS, from 0 to 100), investigating the perceived health.
Chronic illnesses | At the inclusion in the study
  Questions about the presence of chronic illness(es) are asked, along with their duration.
Body Mass Index | At the inclusion in the study
  Calculated with the standard formula (weight/height²)
Feeling of stigma associated with the chronic illness | At the inclusion in the study
  Measured with the Stigma Scale for Chronic Illnesses (Molina et al., 2013), which assesses enacted and internalised stigma. It is composed of 8 items. The responses for each item can be: 1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, and 5 = Always. The raw summed score range is 8-40, with a higher score indicating a higher perceived stigma. Raw scores are then transformed into T-scores (a result of rescaling raw scores into standardized scores with a mean of 50 and a standard deviation of 10).
Satisfaction about health services | At the inclusion in the study
  Investigation of the participant's satisfaction about hospitals, dentists, specialised physician, general practitioners, home care and Solidaris, through 6 questions ranging from 1 (very unsatisfied) to 5 (very satisfied).
Consumption behaviors | At the inclusion in the study
  Tobacco, alcohol, fruits and vegetables consumption are investigated through 5 questions: do you smoke ? / If yes, what do you smoke? / How often do you drink alcohol? / How often do you eat fruits? / How often do you eat vegetables?
Physical activity | At the inclusion in the study
  Investigated through 2 questions: during the last 7 days, how many days did you practice intense physical activity? / during the last 7 days, how many days did you practice moderate physical activity? For each question, answers range from 0 to 7.
Use of the Internet for health purposes | At the inclusion in the study
  Investigated through 1 question: "how often do you use the Internet to search information about your health?". Answers range from 1 (never) to 5 (always).

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - University of Liège, Liège
  - University Hospital of Liege, Liège

IPD SHARING:
Plan to Share IPD: Undecided